CLINICAL TRIAL: NCT06812598
Title: A Clinical Study on the Efficacy of Extended Letermovir Prophylaxis to Prevent CMV Reactivation in High-Risk Chinese Adults Undergoing Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Efficacy of Extended Letermovir Prophylaxis to Prevent CMV Reactivation in High-Risk Chinese Adults Undergoing Allogeneic HSCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SOOCHOW-WXJ-2024-505
Record Dates: First submitted 2025-02-01; First posted 2025-02-06 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-02

CONDITIONS: Cytomegalovirus Infections; CMV
Keywords: Letermovir; Allogeneic Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — letermovir

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): The patient will begin receiving prophylactic treatment with letermovir from day 0 to day 28 post-allo-HSCT, at a dose of 480 mg orally once daily. If administered in combination with cyclosporine, the letermovir dose should be reduced to 240 mg orally once daily. Treatment will continue until 24 weeks post-transplant (approximately 170 days). During hospitalization, the study nurse will distribute the medication to the patient according to the treatment protocol and provide guidance on proper administration. The nurse will ensure the patient adheres to the prescribed dosing schedule and will document both the medication distribution and adherence.
  Interventions: Drug: Letermovir (0-24w）
- Control Group (Other): The patient will begin prophylactic treatment with letermovir from day 0 to day 28 post-allo-HSCT, at a dose of 480 mg orally once daily. If used in combination with cyclosporine, the letermovir dose should be reduced to 240 mg orally once daily. The treatment will continue for up to 14 weeks post-transplant (approximately 100 days). In addition, the usage of the medication will be carefully monitored and documented.
  Interventions: Drug: Letermovir (0-14w）

INTERVENTIONS:
Drug: Letermovir (0-24w） — Patients will begin receiving prophylactic treatment with domestically produced letermovir from day 0 to day 28 post-allo-HSCT, at a dose of 480 mg, administered orally once daily. If used in combination with cyclosporine, the dose should be reduced to 240 mg once daily. The treatment will continue until 24 weeks post-transplant (approximately 170 days).
  Arms: Intervention Group
Drug: Letermovir (0-14w） — Patients will begin receiving prophylactic treatment with domestically produced letermovir from day 0 to day 28 post-allo-HSCT, at a dose of 480 mg, administered orally once daily. If used in combination with cyclosporine, the dose should be reduced to 240 mg once daily. The treatment will continue until 14 weeks post-transplant (approximately 100 days).
  Arms: Control Group

SUMMARY:
After allogeneic hematopoietic stem cell transplantation (allo-HSCT), recipients are immunocompromised and at increased risk of complications, including cytomegalovirus (CMV) infection. International clinical guidelines for the management of CMV infection post-allo-HSCT recommend three main strategies: minimizing infection risk, prevention, and preemptive therapy. However, traditional antiviral agents have not been approved for CMV prophylaxis in allo-HSCT recipients and are associated with significant adverse effects and the development of resistance, leaving the CMV prevention needs of this patient population unmet. Recent studies have demonstrated that letermovir prevents potent and highly specific antiviral activity against CMV, and it has been approved for CMV prophylaxis within the first 100 days post-allo-HSCT. Furthermore, evidence suggests that extending letermovir administration up to 28 weeks further reduces the risk of CMV infection in the later post-transplant period without increasing drug-related mortality. In China, the post-allo-HSCT CMV prevention strategy faces challenges such as limited treatment options, unclear guideline recommendations, non-standardized drug usage in certain medical institutions, and insufficient monitoring. This study aims to provide robust, evidence-based support for the use of letermovir in high-risk CMV reactivation among adult allo-HSCT recipients, thereby broadening clinical treatment choices.

DETAILED DESCRIPTION:
CMV late-onset infections following the discontinuation of letermovir have been reported in numerous clinical studies. During this period, transplant recipients remain in the critical phase of immune reconstitution, and further reducing the occurrence of CMV late-onset infections is crucial for improving transplant outcomes. International data have shown that extending the duration of letermovir prophylaxis can further reduce the risk of CMV infection.

In high-risk populations for CMV reactivation and recurrence, the risk of CMV viremia remains elevated even beyond 100 days post-transplant, with incidence rates ranging from 36% to 54%. Consequently, clinical guidelines recommend extending prophylaxis duration, monitoring periods, and shortening the intervals between tests for these high-risk groups. The Chinese Expert Consensus on the Management of CMV Infection in Allogeneic Hematopoietic Stem Cell Transplantation (2022 Edition) suggests that for high-risk populations, particularly those with acute or chronic GVHD, consideration should be given to extending the treatment course or reinitiating CMV reactivation prevention until immunosuppressive therapy is reduced.

Currently, in China, there are no prospective clinical studies or high-level evidence regarding the extension of prophylactic therapy to reduce CMV late-onset infections in adult allo-HSCT recipients at high risk for CMV reactivation. This study aims to investigate the efficacy and safety of extending letermovir prophylaxis from week 14 to week 24 post-HSCT in patients at high risk of CMV reactivation, thereby offering additional therapeutic options for these patients.

ELIGIBILITY:
Inclusion Criteria:

1. The patients have decided to undergo an initial allogeneic hematopoietic stem cell transplantation (allo-HSCT).
2. The patients are ≥18 years old.
3. The patients are CMV seropositive prior to transplantation.
4. The patients have at least one high-risk factor for CMV reactivation, including:

(1) Haploidentical transplantation, HLA-mismatched transplantation, or unrelated donor transplantation.

(2) The primary source of stem cells is cord blood. (3) A conditioning regimen including total body irradiation (TBI). (4) A GVHD prophylaxis regimen containing alemtuzumab or high-dose anti-thymocyte globulin (ATG).

5. The patients are able to comply with the study visit schedule, understand and agree to adhere to all protocol requirements, and have voluntarily signed the informed consent form to participate in the study.

6. The patients have no plans for reproduction from the date of consent until 90 days after the last dose of the study treatment.

Exclusion Criteria:

1. Patients who have previously received allogeneic hematopoietic stem cell transplantation (allo-HSCT).
2. Patients with evidence of CMV viremia at any time prior to enrollment.
3. Patients with a history of CMV end-organ disease within 6 months prior to enrollment.
4. Patients with suspected or known allergy to letermovir or any active or inactive components of similar drugs.
5. Patients with severe hepatic impairment (defined as Child-Pugh Class C).
6. Patients with end-stage renal disease with a creatinine clearance < 10 mL/min.
7. Patients requiring mechanical ventilation or experiencing hemodynamic instability at the time of enrollment.
8. Patients who received any investigational drug therapy within 28 days prior to enrollment.
9. Patients who received or plan to receive any of the following treatments within 28 days prior to enrollment or during the study: cidofovir, CMV immune globulin, or any experimental CMV antiviral drugs/biological therapies.
10. Patients who previously participated or are currently participating in any study involving a CMV vaccine or other CMV investigational drugs, or who plan to participate in such studies during this trial.
11. Patients who are pregnant or breastfeeding at the time of enrollment or planning to become pregnant within 90 days after the last dose of study medication.
12. Patients who test positive for human immunodeficiency virus antibodies (HIV-Ab) at any time prior to randomization, or who test positive for hepatitis C virus antibodies (HCV-Ab) with detectable HCV RNA, or for hepatitis B surface antigen (HBsAg) within 90 days prior to randomization. Laboratory testing for HIV, HBV, or HCV is allowed using locally acceptable methods.
13. Patients with active solid malignancies, except for localized basal cell or squamous cell carcinoma of the skin or a condition currently under treatment (e.g., lymphoma).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of clinically significant CMV infection (csCMVi) within 24 weeks post-transplant | within 24 weeks following HSCT
  csCMVi: the occurrence of CMV disease or CMV viremia requiring preemptive therapy

SECONDARY OUTCOMES:
Incidence of resistant or refractory CMV infection within 24 weeks post-transplant | within 24 weeks following HSCT
  Refractory CMV viremia: CMV viral load remains unchanged or increases after 2 weeks of appropriate anti-CMV treatment. Refractory CMV disease: Symptoms or signs of CMV disease show no improvement or continue to progress after 2 weeks of appropriate anti-CMV treatment.
Time to initiation of preemptive therapy and duration of treatment for CMV infection within 24 weeks post-transplant | within 24 weeks following HSCT
  Preemptive Therapy for CMV: A treatment strategy where antiviral medications are administered early, based on the detection of CMV reactivation (e.g., through viral load monitoring) before symptoms or disease develop, to prevent the progression to CMV disease.
Incidence and severity of acute graft-versus-host disease (GVHD) within 100 days post-transplant | within 100 days following HSCT
  Acute GVHD: A complication that occurs shortly after allogeneic stem cell transplantation, where the donor's immune cells attack the recipient's tissues, typically affecting the skin, liver, and gastrointestinal tract. It usually develops within the first 100 days post-transplant and can range from mild to severe.
Incidence and severity of chronic GVHD within 24 weeks post-transplant | within 24 weeks following HSCT
  Chronic GVHD: A long-term complication following allogeneic stem cell transplantation, where the donor's immune cells attack the recipient's healthy tissues, affecting organs such as the skin, liver, lungs, and eyes. It can range from mild to severe and may require prolonged immunosuppressive therapy.
Incidence and severity of all adverse events (AEs) within 24 weeks post-transplant | within 24 weeks following HSCT
  Adverse Events (AEs) with letermovir: Refers to any unwanted or harmful effects experienced by patients using letermovir, such as nausea, vomiting, diarrhea, headaches, or elevated liver enzymes. These events can vary in severity and may or may not be related to the medication.
CMV disease-related mortality within 24 weeks post-transplant | within 24 weeks following HSCT
  CMV disease-related mortality: Refers to deaths directly caused by complications of CMV (cytomegalovirus) infection, such as CMV viremia, organ damage, or CMV-related immunosuppression, leading to fatal outcomes.
All-cause mortality and non-relapse mortality within 24 weeks post-transplant | within 24 weeks following HSCT
  All-cause mortality: Refers to deaths from any cause, including disease relapse, treatment complications, or unrelated factors, providing an overall measure of survival. Non-Relapse Mortality (NRM): Refers to deaths unrelated to disease relapse or progression, typically caused by treatment complications such as infections, organ failure, or graft-versus-host disease (GVHD).
  Non-relapse mortality (NRM): Refers to deaths unrelated to disease relapse or progression, typically caused by treatment complications such as infections, organ failure, or graft-versus-host disease (GVHD).

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojin Wu, Prof., Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- Hematology Department, The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China